CLINICAL TRIAL: NCT02500433
Title: Use of a Low Cost Videogame Console in Children With Cerebral Palsy in a School Environment
Brief Title: Virtual Reality in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Laura Luna, PhD, Universidad Rey Juan Carlos
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VR CHILDREN 2015
Record Dates: First submitted 2015-06-09; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; child; rehabilitation; video games; virtual reality.
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device: Kinect-Xbox360TM (Experimental): Based around a webcam-style add-on peripheral for the Xbox 360 console, it enables users to control and interact with the Xbox 360 without the need to touch a game controller, through a natural user interface using gestures and spoken commands. Participants were asked to practice 30 minutes per day, 2 days per week for 2 months, added to their conventional treatment. The games used were Kinect Sports ITM, Kinect Joy RideTM and Kinect Disneyland AdventuresTM and involved balance and trunk movements, general and visual-manual coordination and limb tasks. Each subject followed instructions on the screen with the help of his physiotherapist, with points awarded based on degree and speed of movement and level of difficulty.
  Participants were initially exposed to the games in an hour introductory session, 2 weeks before the study began. All the sessions were supervised by physiotherapist.
  Interventions: Other: Device: Kinect-Xbox 360TM
- Conventional therapy (Other): Conventional therapy was based on neurodevelopment treatment, psychomotor activities and kinesiotherapy during one month, twice per week, with 30 minutes per session.
  The treatment includes: active and passive kinesitherapy, muscle and tendons stretching, training of gait and deambulation, such as coordination and handling.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: Device: Kinect-Xbox 360TM — Based around a webcam-style add-on peripheral for the Xbox 360 console, it enables users to control and interact with the Xbox 360 without the need to touch a game controller, through a natural user interface using gestures and spoken commands. Participants were asked to practice 30 minutes per day, 2 days per week for 2 months, added to their conventional treatment. The games used were Kinect Sports ITM, Kinect Joy RideTM and Kinect Disneyland AdventuresTM and involved balance and trunk movements, general and visual-manual coordination and limb tasks. Each subject followed instructions on the screen with the help of his physiotherapist, with points awarded based on degree and speed of movement and level of difficulty.
  Arms: Device: Kinect-Xbox360TM
Other: Conventional therapy
  Arms: Conventional therapy

SUMMARY:
OBJECTIVE: To investigate whether VR videogames plus conventional therapy improves motor control compared with conventional therapy in children with cerebral palsy (CP).

METHODS: Thirty participants with CP were included. A baseline (A0), a post-conventional intervention (A1), a post-experimental treatment (A2) and a two-month follow-up (A3) assessment were performed. Experimental intervention was based on videogames treatment (Kinect-Kbox360TM) added to their conventional physiotherapy. Motor and the process skills were evaluated by the Assessment of Motor and Process Skills (AMPS); balance by the Pediatric Reach test (PRT); gait speed by the 10-meters walk test (10MW); and running and jumping capacity by the Gross Motor Function Measure (GMFM).

DETAILED DESCRIPTION:
Thirty participants were recruited, seventeen were boys and thirteen were girls, with a mean age of 8.41 years (SD 2.55).

The inclusion and exclusion criteria Children were recruited from Public Schools of Madrid (Spain) and they were classified according to their Gross Motor Function Classification System (GMFCS) level.

The inclusion criteria were a diagnostic of mild-moderate hemiplegic and diplegic CP, age between four to eleven years and receive physiotherapy treatment in the public school related with this project. The exclusion criteria were not have visual impairments, severe cognitive disability, surgical intervention in the year before study onset, botulinum injections in the six months before study onset and non-controlled epilepsy. Six participants were classified as GMFCS level I and twenty-four was level II, all with spastic involvement.

All were receiving physiotherapy at the time of enrollment by the same therapist. All children were enrolled in age-appropriate classes in regular public schools; 100% did receive some extra help for mild learning issues.

Statistical Analyses:

We used a repeated measures analysis of variance (ANOVA) to assess differences among the four assessments in each of the variables, using paired t-test with Bonferroni correction when a significant effect was detected. We performed all the analysis by The Statistical Package for Social Sciences (SPSS 19.0 Version).The statistical analysis was conducted at a 95% confidence level. A p value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of mild-moderate hemiplegic.
* Diplegic cerebral palsy.
* Age between four to eleven years.
* Receive physiotherapy treatment in the public.
* School related with this project

Exclusion Criteria:

* Not Have Visual Impairments.
* Severe Cognitive Disability.
* Surgical Intervention In The Year Before Study Onset.
* Botulinum Injections In The Six Months Before Study Onset.
* Non-Controlled Epilepsy.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Motor and Process Skills (AMPS) | 60 minutes
  Observational assessment used to measure the quality of a person's activities of daily living (ADL). The person performs each prioritized and self-chosen ADL task in a familiar environment and the way he or she usually does it. After completion of each AMPS task observation, the occupational therapist scores the person's quality of performance on each of 16 ADL motor and 20 ADL process items according to the standardized criteria in the AMPS manual. Each task performance observed is scored separately and each ADL skill is rated using a 4-point ordinal scale. Once the evaluation is complete, the therapist enters the raw scores for each ADL task observed into the AMPS software. The AMPS software is then used to perform many-facet Rasch analyses of the person's ordinal raw items scores and generate linear quality of ADL task performance measures.
10-meters walk test (10MW) | 15 minutes
  participants positioned their toes behind the start line and were instructed to walk at their comfortable speed and continue down the corridor until told to stop. Timing began the moment the participant initiated a step and ended when the leading foot crossed the finish line.
Pediatric Reach test (PRT) | 5 minutes
  is a valid and reliable measure with potential for use with children. Children were instructed to lean forward with their arms, moving at their ankles only, as far as possible without lifting their heels off the ground, and to maintain that position for three seconds. The average in centimeters of the three arms reach trials was used.
Gross Motor Function Measure (GMFM). | 45 minutes
  The GMFM is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with CP, is the standard outcome assessment tool for functional intervention in CP. For this paper, standing and gait, running and jumping scales were used.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Luna, PhD, Principal Investigator — Universidad Rey Juna Carlos